CLINICAL TRIAL: NCT05572008
Title: Investigating Protein Nutrition in Paediatric Crohn's Disease
Brief Title: ProteIn Nutrition in Crohn's Disease
Acronym: PINC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 297431
Record Dates: First submitted 2022-09-13; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease (CD); Muscle Protein Synthesis; Muscle Protein Breakdown; Magnetic Resonance Imaging (MRI); Amino Acids (AAs); Essential Amino Acid (EAA)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paediatric Crohn's disease (Experimental): CD young population (ages 12-17 years) - N=20
  Interventions: Behavioral: Protein nutrition in paediatric Crohn's disease
- Healthy volunteers (Active Comparator): Age-, BMI- and gender-matched healthy volunteers (HV) - N=20
  Interventions: Behavioral: Protein nutrition in paediatric Crohn's disease

INTERVENTIONS:
Behavioral: Protein nutrition in paediatric Crohn's disease — All participants (N = 40) will undergo the same study procedures:
  Eating behaviour questionnaire(s) completion Duration: 5 minutes Frequency 2 Dietary intake data via online computerised recall Duration: 60 minutes Frequency: 3 Collection of blood sample via venepuncture Duration: 15 minutes Frequency 1 Strength Tests Duration: 30 minutes Frequency: 1
  Half the participants (N = 20) will return for two more visits and will undergo the following procedures:
  MRI Scan Duration: 30 minutes Frequency: 1 Consumption of intrinsically labelled protein Duration: 15 minutes Frequency: 1 Insertion of cannulae into hand Duration: 15 minutes Frequency: 1 Collection of blood sample via cannulae (for protein digestion and inflammatory markers and study endpoints outlined below) Duration: 1 minute Frequency: 17

SUMMARY:
Muscles are essential for good quality of life. The investigators have shown that when children with Crohn's disease eat protein, only very little of it enters the muscles, leading to poor muscle growth and fatigue. The investigators want to find the reasons for this. The investigators will recruit 20 Crohn's disease patients and a matched group of healthy kids. The investigators will measure:

* Daily food intake and muscle strength.
* Protein absorption by giving our participants a milk protein test drink and take regular blood samples after.
* Muscle mass with MRI. This study will help understand how protein is handled in these patients.

DETAILED DESCRIPTION:
Muscle mass is maintained through the daily balance of muscle protein synthesis (MPS) and muscle protein breakdown (MPB), with the essential amino acid (EAA) components of a meal and muscle contraction being the primary stimulators of MPS. Adult patients with active CD ingest considerably less daily protein intake than age- BMI- matched healthy controls [CD, 70.3 g ± 6.1; HV, 92.6 g ± 7.8, p = 0.03]. Similar observations may be true for children with inactive CD where protein intake is lower with 79 ± 5g/day reported in CD and 90 ± 10g/day reported in HV. In male paediatric patients with long term CD, muscle metabolism is perturbed by a negative branched chain amino acid balance in the forearm. CD may have a significant effect on protein digestion and absorption, blunting the MPS response to feeding, leading to a chronic muscle mass reduction that may persist even when in remission.

The essential amino acid (EAA) components of a protein-meal are crucial for the stimulation of muscle protein synthesis (MPS) and we have shown of all the EAA, leucine plays a key role in driving MPS. Low serum levels EAA/leucine have been reported in adult CD but their role in the aetiology of sarcopenia in paediatric CD is unknown. Further, how CD affects the protein digestion/absorption and how this contributes to low EAA/leucine remains unclear. Recent advances in stable isotope tracer techniques now enable a more accurate determination of protein digestibility. By following the appearance of intrinsically labelled AAs into the blood upon digestion of the intrinsically labelled protein, alongside the appearance of label-free AAs, protein digestibility can be accurately determined.

Main aims: To accurately measure protein intake and fasting plasma EAA and non-EAA in paediatric CD. The investigators will use an intrinsically labelled protein milk to investigate protein digestion and absorption and link these findings to whole body muscle mass as measured through MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-17 years
2. BMI <30 kg/m2 (all)
3. **Documented diagnosis of CD previously confirmed by endoscopy and histology at least 6 months prior to enrolment (CD group only)
4. **Stable CD defined as no change in medication in the last 3 months (including corticosteroids) and no CD-related surgical intervention in the last 6 months (CD group only)
5. Able to participate fully in all aspects of the clinical trial (all)
6. Written informed consent obtained and documented (all) **n/a to HV's

Exclusion Criteria:

1. A current diagnosis of UC, indeterminate colitis or microscopic colitis
2. A diagnosis of short-bowel syndrome
3. Serious underlying disease other than **CD that, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study
4. Contraindications for MRI scanning e.g. pacemaker
5. Dairy intolerance/milk protein allergy
6. Non-English speakers **n/a to HV's

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-12-28 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
Assess protein intake | 15 minutes/ history diary intake
  Detailed 3-days protein intake via Intake24 online questionnaire

SECONDARY OUTCOMES:
Assess calories, carbohydrate, fat and micronutrient intake | 15 minutes/ history diary intake
  Detailed 3-day calorie, carbohydrate, fat and micronutrient intake via Intake24 online questionnaire
Assess eating behaviour | 10 minutes
  Child Eating Behaviour, (CEBQ) questionnaire
Assess eating behaviour | 10 minutes
  Child Tree-Factor Eating Questionnaire (CTFEQr17) questionnaire
Post-prandial protein digestibility | 360 minutes
  Postprandial plasma AA appearance/digestibility via collection of blood sample
Assess body composition | 30 minutes
  Whole-body muscle mass using 3T
Assess body composition | Assess body composition
  Whole-body muscle mass using 3T
Measure serum inflammatory cytokines | 15 minutes
  Serum key cytokines and hormones: IL-1, IL-6, IL-10, IL-15, TNF, GH, IGF-1, testosterone
Quantify muscle strength | 30 minutes
  Muscle strength will be assessed via maximal forearm contractions using a handgrip dynamometer
Assess body composition | 30 minutes
  Intra-myocellular and extra-myocellular lipid content using 3T

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Moran, PhD, Principal Investigator — University of Nottingham; Kostas Tsintzas, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, B Floor, Medical school, Queens Medical centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The samples provided by my child and the information gathered about my child can be stored by the University of Nottingham at the Research Tissue Bank (DI William Dunn-Licence Number 12265), for possible use in future studies
Supporting Information: Study Protocol, ICF
Time Frame: 7 years

REFERENCES:
- [Background] Schneider SM, Al-Jaouni R, Filippi J, Wiroth JB, Zeanandin G, Arab K, Hebuterne X. Sarcopenia is prevalent in patients with Crohn's disease in clinical remission. Inflamm Bowel Dis. 2008 Nov;14(11):1562-8. doi: 10.1002/ibd.20504. PMID 18478564
- [Background] van Langenberg DR, Della Gatta P, Hill B, Zacharewicz E, Gibson PR, Russell AP. Delving into disability in Crohn's disease: dysregulation of molecular pathways may explain skeletal muscle loss in Crohn's disease. J Crohns Colitis. 2014 Jul;8(7):626-34. doi: 10.1016/j.crohns.2013.11.024. Epub 2013 Dec 13. PMID 24332699
- [Background] Gassull MA, Cabre E. Nutrition in inflammatory bowel disease. Curr Opin Clin Nutr Metab Care. 2001 Nov;4(6):561-9. doi: 10.1097/00075197-200111000-00018. PMID 11706295
- [Background] Filippi J, Al-Jaouni R, Wiroth JB, Hebuterne X, Schneider SM. Nutritional deficiencies in patients with Crohn's disease in remission. Inflamm Bowel Dis. 2006 Mar;12(3):185-91. doi: 10.1097/01.MIB.0000206541.15963.c3. PMID 16534419
- [Background] Lochs H, Dejong C, Hammarqvist F, Hebuterne X, Leon-Sanz M, Schutz T, van Gemert W, van Gossum A, Valentini L; DGEM (German Society for Nutritional Medicine); Lubke H, Bischoff S, Engelmann N, Thul P; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Gastroenterology. Clin Nutr. 2006 Apr;25(2):260-74. doi: 10.1016/j.clnu.2006.01.007. Epub 2006 May 15. PMID 16698129
- [Background] Wardle RA, Thapaliya G, Nowak A, Radford S, Dalton M, Finlayson G, Moran GW. An Examination of Appetite and Disordered Eating in Active Crohn's Disease. J Crohns Colitis. 2018 Jun 28;12(7):819-825. doi: 10.1093/ecco-jcc/jjy041. PMID 29617753
- [Background] Davies A, Nixon A, Muhammed R, Tsintzas K, Kirkham S, Stephens FB, Moran GW. Reduced skeletal muscle protein balance in paediatric Crohn's disease. Clin Nutr. 2020 Apr;39(4):1250-1257. doi: 10.1016/j.clnu.2019.05.017. Epub 2019 May 25. PMID 31178247
- [Background] Khalaf A, Hoad CL, Menys A, Nowak A, Radford S, Taylor SA, Latief K, Lingaya M, Falcone Y, Singh G, Spiller RC, Gowland PA, Marciani L, Moran GW. Gastrointestinal peptides and small-bowel hypomotility are possible causes for fasting and postprandial symptoms in active Crohn's disease. Am J Clin Nutr. 2020 Jan 1;111(1):131-140. doi: 10.1093/ajcn/nqz240. PMID 31557279
- [Background] Hisamatsu T, Okamoto S, Hashimoto M, Muramatsu T, Andou A, Uo M, Kitazume MT, Matsuoka K, Yajima T, Inoue N, Kanai T, Ogata H, Iwao Y, Yamakado M, Sakai R, Ono N, Ando T, Suzuki M, Hibi T. Novel, objective, multivariate biomarkers composed of plasma amino acid profiles for the diagnosis and assessment of inflammatory bowel disease. PLoS One. 2012;7(1):e31131. doi: 10.1371/journal.pone.0031131. Epub 2012 Jan 31. PMID 22303484
- [Background] Moughan PJ, Wolfe RR. Determination of Dietary Amino Acid Digestibility in Humans. J Nutr. 2019 Dec 1;149(12):2101-2109. doi: 10.1093/jn/nxz211. PMID 31529051
- [Background] Koopman R, Walrand S, Beelen M, Gijsen AP, Kies AK, Boirie Y, Saris WH, van Loon LJ. Dietary protein digestion and absorption rates and the subsequent postprandial muscle protein synthetic response do not differ between young and elderly men. J Nutr. 2009 Sep;139(9):1707-13. doi: 10.3945/jn.109.109173. Epub 2009 Jul 22. PMID 19625697
- [Background] Tsintzas K, Jones R, Pabla P, Mallinson J, Barrett DA, Kim DH, Cooper S, Davies A, Taylor T, Chee C, Gaffney C, van Loon LJC, Stephens FB. Effect of acute and short-term dietary fat ingestion on postprandial skeletal muscle protein synthesis rates in middle-aged, overweight, and obese men. Am J Physiol Endocrinol Metab. 2020 Mar 1;318(3):E417-E429. doi: 10.1152/ajpendo.00344.2019. Epub 2020 Jan 7. PMID 31910028
- [Background] Koopman R, Crombach N, Gijsen AP, Walrand S, Fauquant J, Kies AK, Lemosquet S, Saris WH, Boirie Y, van Loon LJ. Ingestion of a protein hydrolysate is accompanied by an accelerated in vivo digestion and absorption rate when compared with its intact protein. Am J Clin Nutr. 2009 Jul;90(1):106-15. doi: 10.3945/ajcn.2009.27474. Epub 2009 May 27. PMID 19474134
- [Background] Boirie Y, Fauquant J, Rulquin H, Maubois JL, Beaufrere B. Production of large amounts of [13C]leucine-enriched milk proteins by lactating cows. J Nutr. 1995 Jan;125(1):92-8. doi: 10.1093/jn/125.1.92. PMID 7815181
- [Background] Bradley J, Simpson E, Poliakov I, Matthews JN, Olivier P, Adamson AJ, Foster E. Comparison of INTAKE24 (an Online 24-h Dietary Recall Tool) with Interviewer-Led 24-h Recall in 11-24 Year-Old. Nutrients. 2016 Jun 9;8(6):358. doi: 10.3390/nu8060358. PMID 27294952
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Bryant EJ, Thivel D, Chaput JP, Drapeau V, Blundell JE, King NA. Development and validation of the Child Three-Factor Eating Questionnaire (CTFEQr17). Public Health Nutr. 2018 Oct;21(14):2558-2567. doi: 10.1017/S1368980018001210. Epub 2018 May 15. PMID 29759100
- [Background] Gallen IW, Macdonald IA. Effect of two methods of hand heating on body temperature, forearm blood flow, and deep venous oxygen saturation. Am J Physiol. 1990 Nov;259(5 Pt 1):E639-43. doi: 10.1152/ajpendo.1990.259.5.E639. PMID 2240202
- [Background] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845